CLINICAL TRIAL: NCT00005927
Title: Clinical and Molecular Analysis of ACTH-Independent Steroid Hormone Production in Adrenocortical Tissue
Brief Title: Study of Adrenal Gland Tumors
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000160; 00-CH-0160
Record Dates: First submitted 2000-06-28; First posted 2000-06-29 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-12-10

CONDITIONS: Adrenal Gland Neoplasm
Keywords: Macronodular Adrenals; Cushing's Syndrome; Adrenal Gland; Natural History
MeSH Terms: conditions — Adrenal Gland Neoplasms; Cushing Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hyperaldosteronism and cushing participants: Subjects with Hyperaldosteronism and cushing. Adults, pediatric subjects and family members (DNA collection only for family members).

SUMMARY:
The adrenal glands, located atop the kidneys, normally produce several types of hormones. Tumors of these glands may or may not secrete hormones. It is not known what causes these tumors or why some secrete hormones and others do not. Some of the tumors are benign and confined to the adrenal gland, and others are malignant (cancerous), and can spread to other parts of the body. This study will investigate how adrenal gland tumors develop, why some secrete steroid hormones and others do not, and why some are benign and others malignant.

Patients between 3 and 70 years old with a known or suspected adrenal gland tumor may be eligible for this study. Participants will be hospitalized for 7 to 10 days for various tests and procedures that may include the following:

1. Medical history and physical examination, including body measurements, as appropriate. Children and adolescents will have Tanner staging, including examination of the genitals, to determine the extent of sexual maturity.
2. 24-hour urine collection to measure hormones in the urine.
3. Imaging studies, including magnetic resonance imaging (MRI) of the brain, computed tomography (CT) and other X-ray studies.
4. Blood tests to see if the tumor secretes hormones in response to specific stimuli, including exercise, food, and various hormones. The hormones are given through an intravenous catheter, or IV a thin plastic tube inserted into an arm vein. After the stimulus, blood is drawn through the same IV every 30 minutes for up to 3 hours to measure hormone levels. Based on the results of these tests, some patients may have additional blood tests to check hormone response to special foods, an IV salt solution, or other hormones or drugs given either IV or by mouth (in pill form).
5. Photographs to document the effects on the body of abnormal hormone secretion from the adrenal tumor.
6. Small samples of blood and tumor tissue for research and DNA (genetic) analysis.

A discussion of treatment options will be based on the results of tests. If surgery to remove the tumor is recommended, the procedure can be done at NIH under this study protocol. If a malignant tumor is found that cannot be treated surgically, chemotherapy or radiation therapy may be recommended. These options are not offered under this protocol, but may be available under a different NIH study (for example, at the National Cancer Institute). Referrals will be made at the patient s request.

Patients who had surgery may be followed at the NIH outpatient clinic for 1 year after surgery. Patients with certain types of tumors may continue to be followed at NIH once a year for up to 5 years.

A registry of study participants will be created to keep records and correlate medical histories with tissues kept at NIH. The registry will also be used to inform participants of research studies they may be interested in. No individuals or organizations outside of NIH will have access to the registry.

DETAILED DESCRIPTION:
The adrenal glands are the major source in the body of the steroid hormones. In normal physiology, the pituitary hormone ACTH regulates the secretion of glucocorticoids, while the secretion of mineralocorticoids such as aldosterone is controlled by the renin-angiotensin system. In addition to these two classes of steroids, the adrenal gland secretes lesser amounts of intermediate metabolites as well as dehydroepiandrosterone (DHEA) and its sulfated product (DHEAS) and androstenedione, testosterone, estrogen, and estrone. Dysregulated secretion of any of these hormones can be caused by sporadic adrenocortical adenomas or carcinomas, with the development of specific clinical syndromes depending on the identity of the hormones secreted. In at least a subset of cortisol-producing adrenocortical neoplasms, the presence of ectopic or abnormal receptors has been described, resulting in the regulation of cortisol and/or aldosterone by non-physiologic stimuli. The present study will serve as a mechanism to investigate individuals with steroid hormone-secreting adrenocortical tumors of all types for the purpose of identifying hereditary, congenital, or acquired defects leading not only to hormone oversecretion, but also to tumor formation. One of the first goals of the study was (until very recently) to examine the prevalence of ectopic receptor expression in cortisol- and/or aldosterone- hormone secreting adrenocortical tumors. This led to the understanding of the ontogeny of these tumors and the development of novel therapeutic strategies (e.g., receptor antagonists) to control hormone oversecretion. We currently use this information for the evaluation and treatment of our patients. An important research goal of the study is to identify novel genetic defects leading to tumors of the adrenal gland. This is done through a set of methods, from sequencing of the collected DNA to analysis of the expression of large sets of genes using gene array/gene chip analysis. This information may help to identify patients who would benefit from more aggressive intervention strategies, especially those with potentially malignant tumors. This study also provides the patient cohort necessary for the establishment of a bank of tissues of varying tumors of the adrenal cortex, which may serve in the future as an experimental resource to test new diagnostic and therapeutic methods. Finally, an important and more recent goal of this study is to investigate the effects of excess aldosterone on renal, cardiac, metabolic, and bone systems in patients with primary hyperaldosteronism, an important subgroup of patients with adrenocortical tumors. Patients with hyperaldosetronism have not been studied with the same rigor as patients with hypercortisolism in the past; this study aims at investigating the relative contribution of hyperaldosteronism in the etiopathogenesis of a number of clinical problems in patients with adrenocortical lesions and hypertension.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients are adults or children with evidence for the existence of a tumor of the adrenal glands, as indicated by previously obtained imaging studies and/or biochemical investigation of hormonal secretion. This condition is meant to include the possibility of individuals with "sub-clinical" hormone secretion syndromes, which may be detectable at the biochemical level even in the absence of frank clinical signs/symptoms.

All eligible patients are invited to participate in this protocol, regardless of sex, race or ethnic origin. All populations appear at risk for adrenal tumors, and therefore the subject population can include Native Americans, Asian/Pacific Islanders, Caucasian, Hispanic, and Black individuals. Patients will be accepted for evaluation based on referral from clinicians, or may be self-referred, if they can provide evidence supportive of the diagnosis of hormone over-secretion.

Patients must be willing to return to the NIH for follow-up evaluation.

Patients may withdraw from the study at any time.

EXCLUSION CRITERIA:

1. Children less than 3 years old will be excluded from the protocol because of the limited resources available at the NIH for the care of infants of this age.
2. Individuals over the age of 70 years of age will be excluded because of the possibility of comorbidities that may significantly affect appropriate initial work-up and post-operative management. In addition, research data may be compromised by the inability to interpret data collected from patients over the age of 70 years that may be on multiple medications for a variety for reasons.
3. Women who are pregnant or nursing will be excluded from the hyperaldosteronism arm of the protocol. Women with adrenal tumors secreting cortisol or other adrenal hormones may benefit clinically from evaluation and treatment of their tumor, and will be considered for enrollment when clinically indicated.
4. Individuals whose medical status will not allow them, for safety reasons, to participate in the provocative testing or who have unacceptably high risk for surgical morbidity and mortality will be excluded from the protocol, as they will not be able to participate profitably in the research aspects of this protocol.
5. Individuals found to have an known inherited syndrome as the cause for hormone oversecretion will be excluded from participation in this protocol, as the mechanisms of hormone oversecretion and tumorigenesis is likely to be distinct in these individuals. Specific examples of syndromes to may be excluded from this protocol include individuals with Carney Complex, McCune-Albright syndrome, and MEN-1. If inquiries are received from such patients, they will be referred to the appropriate ongoing protocols, if possible.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Research subjects who present with Adrenal adenoma, adrenal carcinoma, Cushing syndrome, virilizing adrenals tumor, feminizing adrenal tumor, massive macronodular adrenocortical disease, ACTH-independent macronodular adrenal hyperplasia
Sampling Method: Non-Probability Sample
Enrollment: 690 (Actual)
Dates: Start 2002-07-01 (Actual)

PRIMARY OUTCOMES:
To study the contribution of ectopic/abnormal membrane hormone receptor expression in the adrenal gland to the pathogenesis of primary adrenocortical hormone over-secretion syndromes | This is an ongoing project
  -to define the germline and/or somatic genetic mutations causing ACTH-independent Cushing s syndrome -to define the biochemical functionality of mutations in adrenocortical tumor -to investigate novel therapeutic strategies to control hormone over-secretion of biochemically active adrenal tumors

SECONDARY OUTCOMES:
To investigate the renal, cardiac, metabolic, and bone effects of hyperaldosteronism. To utilize high-density gene array analysis to identify patterns of gene expression that will discriminate between benign and malignant adrenal tumors. | This is an ongoing project
  to investigate co-secretion of other steroids -to investigate cardiac, renal, metabolic and coagulopathic consequences of primary aldosteronism -to investigate the clinical utility of other biomarkers in classifying adrenal disorders

CONTACTS AND LOCATIONS:
Overall Officials: Deborah P Merke, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Torpy DJ, Stratakis CA, Chrousos GP. Hyper- and hypoaldosteronism. Vitam Horm. 1999;57:177-216. doi: 10.1016/s0083-6729(08)60644-5. PMID 10232050
- [Background] Dluhy RG, Lifton RP. Glucocorticoid-remediable aldosteronism. J Clin Endocrinol Metab. 1999 Dec;84(12):4341-4. doi: 10.1210/jcem.84.12.6256. No abstract available. PMID 10599685
- [Background] Torpy DJ, Gordon RD, Lin JP, Huggard PR, Taymans SE, Stowasser M, Chrousos GP, Stratakis CA. Familial hyperaldosteronism type II: description of a large kindred and exclusion of the aldosterone synthase (CYP11B2) gene. J Clin Endocrinol Metab. 1998 Sep;83(9):3214-8. doi: 10.1210/jcem.83.9.5086. PMID 9745430
- [Derived] Hodes A, Meyer J, Lodish MB, Stratakis CA, Zilbermint M. Mini-review of hair cortisol concentration for evaluation of Cushing syndrome. Expert Rev Endocrinol Metab. 2018 Sep;13(5):225-231. doi: 10.1080/17446651.2018.1517043. Epub 2018 Sep 20. PMID 30234410
- [Derived] Angelousi A, Fencl F, Faucz FR, Malikova J, Sumnik Z, Lebl J, Stratakis CA. McCune Albright syndrome and bilateral adrenal hyperplasia: the GNAS mutation may only be present in adrenal tissue. Hormones (Athens). 2015 Jul-Sep;14(3):447-50. doi: 10.14310/horm.2002.1578. PMID 26188235
- [Derived] Neychev V, Steinberg SM, Yang L, Mehta A, Nilubol N, Keil MF, Nieman L, Stratakis CA, Kebebew E. Long-Term Outcome of Bilateral Laparoscopic Adrenalectomy Measured by Disease-Specific Questionnaire in a Unique Group of Patients with Cushing's Syndrome. Ann Surg Oncol. 2015 Dec;22 Suppl 3(Suppl 3):S699-706. doi: 10.1245/s10434-015-4605-1. Epub 2015 May 13. PMID 25968622
- [Derived] Zilbermint M, Xekouki P, Faucz FR, Berthon A, Gkourogianni A, Schernthaner-Reiter MH, Batsis M, Sinaii N, Quezado MM, Merino M, Hodes A, Abraham SB, Libe R, Assie G, Espiard S, Drougat L, Ragazzon B, Davis A, Gebreab SY, Neff R, Kebebew E, Bertherat J, Lodish MB, Stratakis CA. Primary Aldosteronism and ARMC5 Variants. J Clin Endocrinol Metab. 2015 Jun;100(6):E900-9. doi: 10.1210/jc.2014-4167. Epub 2015 Mar 30. PMID 25822102
- [Derived] Keil MF, Graf J, Gokarn N, Stratakis CA. Anthropometric measures and fasting insulin levels in children before and after cure of Cushing syndrome. Clin Nutr. 2012 Jun;31(3):359-63. doi: 10.1016/j.clnu.2011.11.007. Epub 2011 Dec 7. PMID 22154461
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2000-CH-0160.html